CLINICAL TRIAL: NCT01123044
Title: Transplantation of Cultivated Corneal Epithelial Sheet in Patients With Ocular Surface Disease
Acronym: CLET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Head Clinical Trial Unit, Clinical Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 09-01
Record Dates: First submitted 2010-04-22; First posted 2010-05-14 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2010-05

CONDITIONS: Eye Injury
MeSH Terms: conditions — Eye Injuries | interventions — Conservative Treatment; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- corneal stem cell transplant (Experimental)
  Interventions: Biological: conservative
- conservative medical therapy (No Intervention)
  Interventions: Biological: conservative; Procedure: Medical Therapy

INTERVENTIONS:
Biological: conservative — Undergo autologous transplantation of limbal epithelial cells cultured on amniotic membrane
Procedure: Medical Therapy — Under usual care treatment
  Arms: conservative medical therapy

SUMMARY:
The aim of the study is to assess if transplantation of cultivated corneal epithelial stem cells could restore vision in patients with severe ocular surface disorder with a favourable safety profile that warrants further comparative study.

DETAILED DESCRIPTION:
Objectives:

Efficacy:

To determine the efficacy of cultivated corneal epithelial stem cells as a treatment for patients with severe ocular surface disorder.

The corneal limbal epithelial stem cell transplant (CLET) successful outcome will be measured by improvement of vision, maintenance of corneal re-epithelisation with absence of recurrence of surface disease and subjective improvement of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant females between 18 and 75 years of age.
2. Written informed consent obtained from patient or parents/guardian.
3. Patients with unilateral limbal stem deficiency 2-12 months presenting with any of the following

   * Conjunctivalisation
   * Absence of limbal palisades of Vogts
   * Chronic inflammation
   * Persistent or recurrent corneal epithelial defect
4. Patients who had 2-12 months of conservative treatment. * Diagnostic criteria for limbal stem cell deficiency are as follows:

   * Symptoms of decreased vision, redness, watering, photophobia and recurrent attacks of pain
   * Triad of signs: conjunctivalisation, neovascularisation and chronic inflammation
   * Stippled appearance of cunjunctivalised cornea with loss of palisades of Vogt
   * Recurrent and persistent epithelial defects
   * Superficial vascularisation, scarring, thick fibrovascular pannus, ulceration, melting and perforation

Exclusion Criteria:

Patients with any of the following are not eligible for enrollment into the study:

1. Pregnant or nursing woman or women of childbearing potential except if post-menopausal, surgically sterile or using accepted method(s) of birth control or having negative pregnancy test.
2. Participation in any drug trial in which the patient received an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the screening phase of this study.
3. Those persons directly involved in the conduct of the study.
4. Any history of severe infection such as hepatitis, renal, gastrointestinal, endocrine or neurological disease.
5. Evidence of corneal stromal scarring, cataract, macular oedema or scarring, retinal detachment and conjunctival keratinisation
6. Positive for HIV, Hepatitis B, C and VDRL
7. History of Pulmonary tuberculosis, hepatitis B,
8. History of alcohol or substance abuse
9. History of malignancy within previous 5 years
10. History of organ transplant
11. Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Improvement of vision at one week | One week
  The primary efficacy variable will be improved visual acuity Vision will be assessed using ETDRS logMAR visual acuity measurements. An improvement of > 1 line
Improvement of vision at one month | One month
  The primary efficacy variable will be improved visual acuity Vision will be assessed using ETDRS logMAR visual acuity measurements. An improvement of > 1 line
Improvement of vision at three month | Three month
  The primary efficacy variable will be improved visual acuity Vision will be assessed using ETDRS logMAR visual acuity measurements. An improvement of > 1 line
Improvement of vision at six month | Six month
  The primary efficacy variable will be improved visual acuity Vision will be assessed using ETDRS logMAR visual acuity measurements. An improvement of > 1 line
Improvement of vision at nine month | Nine month
  The primary efficacy variable will be improved visual acuity Vision will be assessed using ETDRS logMAR visual acuity measurements. An improvement of > 1 line
Improvement of vision at twelve month | Twelve month
  The primary efficacy variable will be improved visual acuity Vision will be assessed using ETDRS logMAR visual acuity measurements. An improvement of > 1 line

SECONDARY OUTCOMES:
Adverse events reporting, vital signs, and physical examinations.
  To evaluate the safety and tolerability of transplantation of limbal epithelial cells cultured on amniotic membrane for a follow-up period of one year in patients. Safety will be evaluated using adverse events reporting, vital signs, and physical examinations.
Maintenance of corneal re-epithelisation with absence of recurrence of surface disease
Subjective improvement of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur, Malaysia